CLINICAL TRIAL: NCT02592746
Title: A Phase II Randomized Study of Palbociclib in Combination With Exemestane Plus GnRH Versus Capecitabine in Premenopausal Women With Hormone Receptor-Positive Metastatic Breast Cancer
Brief Title: A Study of Palbociclib With Exemestane Plus GnRH Versus Capecitabine in Premenopausal Women With HR+ MBC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, MD, Ph.D, Division of Hematology-Oncology, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-08-042
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; exemestane; Leuprolide; Gonadotropin-Releasing Hormone; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palbociclib + Exemestane + GnRH agonist (Experimental)
  Interventions: Drug: Palbociclib; Drug: Exemestane; Drug: Leuprolide Acetate
- Capecitabine (Active Comparator)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Palbociclib — Palbociclib 125mg, orally once daily on D1 to D21 followed by 7days off
  Other Names: PD-0332991
  Arms: Palbociclib + Exemestane + GnRH agonist
Drug: Exemestane — Exemestane 25mg, orally once daily
  Other Names: FCE-24304
  Arms: Palbociclib + Exemestane + GnRH agonist
Drug: Leuprolide Acetate — Leuprolide Acetate 3.75mg SC q 4weeks
  Other Names: GnRH agonist
  Arms: Palbociclib + Exemestane + GnRH agonist
Drug: Capecitabine — Capecitabine 1,250mg/m2 bid orally form day1 to day 14 q 3weeks
  Other Names: Xeloda
  Arms: Capecitabine

SUMMARY:
Despite recent advances for the treatment of post-menopausal hormone receptor-positive BC, in the last decade there was no major improvement of hormonal therapy specifically for premenopausal metastatic breast cancer. The median age of breast cancer is much younger, and the proportion of young breast cancer (YBC) patients (less than 40) including premenopausal women is much higher, in Asia, including Korea.

Capecitabine, the comparator in this trial, is an orally-administered fluoropyrimidine derivative and has shown high efficacy and low toxicity in metastatic breast cancer patients. Palbociclib is a CDK4/6 inhibitors, in combination with endocrine therapy showed marked advance in hormone receptor-positive MBC in the post-menopausal setting. After a median follow-up of 16.5 months, preliminary results from Part 1 of this Phase 2 trial suggest that the combination of PD-0332991 with letrozole is superior to letrozole alone, and improved objective response and disease control rates (52% vs 32% and 76% vs 47%, respectively) in patients treated with the combination. These remarkable results may contribute to have much benefit with endocrine therapy for premenopausal women. Most importantly, recent PALOMA-3 trial revealed superior results of adding palbociclib to fulvestrant (median PFS 9.2 vs 3.8 months, P<0.001).

Based on these rational backgrounds, the purpose of this phase II study is to assess the safety and the clinical anti-tumor activity of exemestane plus goserelin acetate in combination with palbociclib vs capecitabine in premenopausal hormone receptor-positive advanced breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic breast cancer with measurable or evaluable disease: Patients who have progressed on distant metastatic sites after curative surgery or have stage IV breast cancer at diagnosis
2. Age > 19 years
3. ECOG performance status 0 - 2
4. Patient has HER2-negative breast cancer with IHC and/or FISH (or SISH, CISH) Patient has ER positive and/or PgR positive breast cancer by local laboratory testing
5. Patient is premenopausal. Premenopausal status is defined as either:

   A. Patient had last menstrual period within the last 12 months B. If within three months of tamoxifen (tamoxifen) taking, C. In case of chemotherapy induced amenorrhea, the serum FSH ≤40IU/l
6. A. Patient who have stage IV breast cancer at diagnosis, allow disease that progressed after 1st line chemotherapy. B. Patient who have stage IV breast cancer at diagnosis, allow disease that progressed after tamoxifen or goserelin. C. In case of recur/metastatic breast cancer, allow disease that progressed after 12 month of completion of neo/adjuvant chemotherapy .
7. Urine or serum HCG test must be negative.
8. Adequate bone marrow function (≥ ANC 1,500/ul, ≥ platelet 100,000/ul, ≥ Hemoglobin 9.0 g/dl)
9. Adequate renal function (≤ serum creatinine 1.5 mg/dl or CCr ≥ 50 ml/min)
10. Adequate liver function (≤ serum bilirubin 1.5 mg/dl, ≤ AST/ALT x 3 upper normal limit)
11. Patients who were already established on bisphosphonate therapy may continue on bisphosphonates.
12. Patients agreed to use effective contraception or not of childbearing potential
13. Written informed consent
14. Consent to biomarker analysis.

Exclusion Criteria:

1. Postmenopausal women
2. Serious uncontrolled intercurrent infections
3. Serious intercurrent medical or psychiatric illness, including active cardiac disease
4. Pregnancy or breast feeding
5. Second primary malignancy(except in situ carcinoma of the cervix or adequately treated nonmelanomatous carcinoma of the skin or resected thyroid papillary carcinoma or other malignancy treated at least 5 years previously with no evidence of recurrence)
6. Patients has received previous endocrine treatments such as, aromatase inhibitor, exemestane in the metastatic setting
7. Patients has received previous treatment with CDK 4/6 inhibitors, mTOR inhibitors, PIK3CA inhibitors or capecitabine
8. No symptomatic visceral metastasis
9. Known brain metastases unless treated and stable
10. Clinically significant uncontrolled conditions including, known active hepatitis B or hepatitis C.
11. QTc interval > 480 msec, family or personal history of long or short QT syndrome, or known history of QTc prolongation or Torsade de Pointes.
12. Known positive testing for human immunodeficiency virus or acquired immune deficiency syndrome.
13. Unable to swallow and retain oral medication.
14. Treatment radiotherapy within 4 weeks of the study
15. Use of any investigational drug within 4 weeks of the study
16. Treatment with chemotherapy within 3 weeks or hormone therapy within 2 weeks of the study

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2016-06; Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) in patients with metastatic breast cancer who received palbociclib plus exemestane with goserelin versus capecitabine | 1year

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Ahn HK, Kim JY, Lee KH, Kim GM, Kang SY, Lee KS, Kim JH, Lee KE, Lee MH, Kim HJ, Kim HJ, Koh SJ, Park IH, Sohn J, Kim SB, Ahn JS, Kim S, Cho H, Jung KH, Im SA, Park YH; Korean Cancer Study Group (KCSG) Breast Cancer Committee. Palbociclib plus endocrine therapy versus capecitabine in premenopausal women with hormone receptor-positive, HER2-negative metastatic breast cancer (Young-PEARL): overall survival analysis of a randomised, open-label, phase 2 study. Lancet Oncol. 2025 Mar;26(3):343-354. doi: 10.1016/S1470-2045(25)00006-3. Epub 2025 Feb 17. PMID 39978378
- [Derived] Park YH, Kim TY, Kim GM, Kang SY, Park IH, Kim JH, Lee KE, Ahn HK, Lee MH, Kim HJ, Kim HJ, Lee JI, Koh SJ, Kim JY, Lee KH, Sohn J, Kim SB, Ahn JS, Im YH, Jung KH, Im SA; Korean Cancer Study Group (KCSG). Palbociclib plus exemestane with gonadotropin-releasing hormone agonist versus capecitabine in premenopausal women with hormone receptor-positive, HER2-negative metastatic breast cancer (KCSG-BR15-10): a multicentre, open-label, randomised, phase 2 trial. Lancet Oncol. 2019 Dec;20(12):1750-1759. doi: 10.1016/S1470-2045(19)30565-0. Epub 2019 Oct 24. PMID 31668850